CLINICAL TRIAL: NCT03116217
Title: Multicentre Validation of a Fetal Urine Peptidome-based Classifier to Predict Post-natal Renal Function in Posterior Urethral Valves
Brief Title: Validation of a Fetal Urine Peptidome-based Classifier to Predict Post-natal Renal Function in Posterior Urethral Valves
Acronym: Antenatal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/8805; 2016-A01914-47 (Other: ID-RCB)
Record Dates: First submitted 2017-03-10; First posted 2017-04-17 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Posterior Urethral Valves
Keywords: renal function; post natal; peptidome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validate the use of fetal urine peptidome-analysis and explore amniotic fluid markers for the stratification of fetuses with Posterior Urethral Valve for post-natal renal function.

DETAILED DESCRIPTION:
The ANTENATAL project requires the use of fetal urine as well as post-natal urine, post-natal serum and, possibly, amniotic liquid. We will take an additional tube during the takings collected for routine management of the disease.

The analysis of samples will be carried out in Toulouse at the Institute of Metabolic and Cardiovascular Diseases or with fee-for-service suppliers.

ELIGIBILITY:
Inclusion Criteria:

* male singleton fetus with megabladder associated with urinary tract anomalies with or without dysplastic or hyperechogenic parenchyma detected in a first ultrasound;
* megabladder confirmed in a second ultrasound;
* collection of fetal urine taken during the routine management of the disease for the dosage of ß2-microglobulin;
* written informed consent.

Exclusion Criteria:

* refusal to participate in the study;
* person protected by law.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Mothers (18 years old and more) carrying male fetuses with suspected PUV
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2023-12-26 (Estimated)

PRIMARY OUTCOMES:
Renal/patient survival at 2 years post-natally. | Year 2
  Defined by the need for dialysis or death.

SECONDARY OUTCOMES:
Renal function of the survivors at day 4 and 6 and 12 month post-natally. | Year 1
  This post-natal renal function, estimated via serum cystatin C concentrations, will be analysed centrally in Toulouse to homogenise the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DECRAMER, Pr, Principal Investigator — University Hospital, Toulouse
Locations (29):
- UZ Leuven, Leuven, Belgium
- France (20):
  - CHU Pellegrin-Bordeaux, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Brest
  - Hôpital Femme Mère Enfant-Lyon, Bron
  - CH René-Dubos, Cergy-Pontoise
  - CHU Estaing, Clermont-Ferrand
  - CHU de Grenoble - Hôpital Couple-Enfant - Département de la Génétique, Grenoble
  - CHU de la Timone, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Hôpital mère-enfant pédiatrie, Nantes
  - CHU Lenval, Nice
  - AP-HP - Hôpital Necker Enfants malades, Paris
  - Hôpital Robert-Debré, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes Hôpital Sud, Rennes
  - CHU Hôpitaux de St-Etienne-Hôpital Nord, Saint-Etienne
  - Centre hospitalier universitaire Chu Amiens Salouël Hôpital sud, Salouël
  - Sihcus-Cmco, Schiltigheim
  - Hôpital Bagatelle (Talence) - CHU Pellegrin (Bordeaux), Talence
  - Hôpital Paule de Viguier-Hôpital des enfants- Site Purpan, Toulouse
  - Centre Olympe de Gouges du CHRU de Tours, Tours
- Heidelberg University Hospital, Heidelberg, Germany
- Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico, Milan, Italy
- Netherlands (2):
  - Leiden University Medical Center Dept of prenatal diagnosis and therapy, Leiden, The Netherlands
  - Radboudumc Amalia Children's Hospital, Nijmegen, The Netherlands
- Polish Mothers Memorial Hospital Research Institute, Lodz, Poland
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Hôpital des Enfants Hôpitaux universitaire Genève (HUG), Geneva, Switserland, Switzerland
- FetalMedicine Centre Birmingham Women's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hogan J, Dourthe ME, Blondiaux E, Jouannic JM, Garel C, Ulinski T. Renal outcome in children with antenatal diagnosis of severe CAKUT. Pediatr Nephrol. 2012 Mar;27(3):497-502. doi: 10.1007/s00467-011-2068-6. Epub 2011 Dec 14. PMID 22167562
- [Background] Seeds JW. Diagnostic mid trimester amniocentesis: how safe? Am J Obstet Gynecol. 2004 Aug;191(2):607-15. doi: 10.1016/j.ajog.2004.05.078. PMID 15343248
- [Background] Clark TJ, Martin WL, Divakaran TG, Whittle MJ, Kilby MD, Khan KS. Prenatal bladder drainage in the management of fetal lower urinary tract obstruction: a systematic review and meta-analysis. Obstet Gynecol. 2003 Aug;102(2):367-82. doi: 10.1016/s0029-7844(03)00577-5. PMID 12907115
- [Background] Morris RK, Malin GL, Quinlan-Jones E, Middleton LJ, Hemming K, Burke D, Daniels JP, Khan KS, Deeks J, Kilby MD; Percutaneous vesicoamniotic shunting in Lower Urinary Tract Obstruction (PLUTO) Collaborative Group. Percutaneous vesicoamniotic shunting versus conservative management for fetal lower urinary tract obstruction (PLUTO): a randomised trial. Lancet. 2013 Nov 2;382(9903):1496-506. doi: 10.1016/S0140-6736(13)60992-7. Epub 2013 Aug 14. PMID 23953766
- [Background] Schmoor C, Sauerbrei W, Schumacher M. Sample size considerations for the evaluation of prognostic factors in survival analysis. Stat Med. 2000 Feb 29;19(4):441-52. doi: 10.1002/(sici)1097-0258(20000229)19:43.0.co;2-n. PMID 10694729
- [Background] Lijmer JG, Mol BW, Heisterkamp S, Bonsel GJ, Prins MH, van der Meulen JH, Bossuyt PM. Empirical evidence of design-related bias in studies of diagnostic tests. JAMA. 1999 Sep 15;282(11):1061-6. doi: 10.1001/jama.282.11.1061. PMID 10493205
- [Background] Rutjes AW, Reitsma JB, Di Nisio M, Smidt N, van Rijn JC, Bossuyt PM. Evidence of bias and variation in diagnostic accuracy studies. CMAJ. 2006 Feb 14;174(4):469-76. doi: 10.1503/cmaj.050090. PMID 16477057
- [Background] Donders AR, van der Heijden GJ, Stijnen T, Moons KG. Review: a gentle introduction to imputation of missing values. J Clin Epidemiol. 2006 Oct;59(10):1087-91. doi: 10.1016/j.jclinepi.2006.01.014. Epub 2006 Jul 11. PMID 16980149
- [Background] Klein J, Lacroix C, Caubet C, Siwy J, Zurbig P, Dakna M, Muller F, Breuil B, Stalmach A, Mullen W, Mischak H, Bandin F, Monsarrat B, Bascands JL, Decramer S, Schanstra JP. Fetal urinary peptides to predict postnatal outcome of renal disease in fetuses with posterior urethral valves (PUV). Sci Transl Med. 2013 Aug 14;5(198):198ra106. doi: 10.1126/scitranslmed.3005807. PMID 23946195